CLINICAL TRIAL: NCT02193308
Title: Bioequivalence of 80 mg Telmisartan / 10 mg Amlodipine Fixed Dose Combination Compared With Its Monocomponents in Healthy Male and Female Volunteers. An Open-label, Randomised, Single-dose, Two Sequence, Two-period Crossover Study
Brief Title: Bioequivalence of Telmisartan/Amlodipine Fixed Dose Combination Compared With Its Monocomponents in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.4
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Amlodipine

ARMS (2):
- Telmisartan/Amlodipine FDC (Experimental)
  Interventions: Drug: Telmisartan/Amlodipine FDC
- Telmisartan + Amlodipine mono (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: Amlodipine

INTERVENTIONS:
Drug: Telmisartan/Amlodipine FDC
  Arms: Telmisartan/Amlodipine FDC
Drug: Telmisartan
  Arms: Telmisartan + Amlodipine mono
Drug: Amlodipine
  Arms: Telmisartan + Amlodipine mono

SUMMARY:
To demonstrate the bioequivalence of 80 mg telmisartan / 10 mg amlodipine fixed dose combination (FDC) vs. its monocomponents

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and ≤55 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial (especially unspecific inducing agents like St.John´s wort (Hypericum perforatum) or inhibitors like cimetidine) or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
13. Inability to refrain from smoking during 24 hours prior to dosing and during the trial
14. Alcohol abuse or inability to stop alcoholic beverages for 24 hours prior to dosing and during the trial
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
21. A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hyperkalemia, hypokalemia, family history of Long QT Syndrome)
22. Any history of relevant low blood pressure
23. Supine blood pressure at screening of systolic <110 mm Hg and diastolic <60 mm Hg
24. History of urticaria
25. History of angioneurotic edema
26. Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
27. No adequate contraception during the study and until 1 month of study completion, i.e. implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females, who have not a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
28. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 168 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 168 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 168 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 168 hours after drug administration
λz (terminal rate constant in plasma) | up to 168 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 168 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 168 hours after drug administration
CL/F (apparent clearance of the analyte in plasma after oral administration) | up to 168 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz after oral administration) | up to 168 hours after drug administration
Number of patients with adverse events | up to 65 days
Assessment of tolerability by investigator on a 4-point scale | Day 8 of each trial period